CLINICAL TRIAL: NCT03787537
Title: Assessing Nutritional Status and Nutrient Supply in Hospitalised Patients Undergoing Major Abdominal Surgery of the Gastrointestinal Tract
Brief Title: Nutritional Status and Nutrient Supply in Hospitalised Surgical Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Felix Aigner, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA2/094/17
Record Dates: First submitted 2018-12-07; First posted 2018-12-26 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Gastric Cancer
Keywords: Nutrition; Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective single arm, single center observational study to assess the nutritional status and the nutrient supply during hospitalization for elective gastrointestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective surgery of the upper or lower gastrointestinal tract
* mental and verbal ability to understand, read and write in German language
* written informed consent for study participation

Exclusion Criteria:

* age <18 years
* inadequate ability to be compliant with the study protocol or to complete documentation for the Food frequency questionnaires

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in nutritional status | 24 hours pre-surgery and 7 days after surgery
  Controlling Nutritional Status (CONUT) score will be assessed at baseline and on postoperative day 7

SECONDARY OUTCOMES:
Energy intake | 1 day before surgery, the day of surgery and up to 7 days after surgery
  Dietary intakes are collected by Food Frequency questionnaires and the data are expressed as the kilocalories (kcal) consumed per day
Change in plasma amino acid levels | 24 hours pre-surgery up to 7 days after surgery
  Blood sample analysis
Change in beta-hydroxybutyrate levels | 24 hours pre-surgery up to 7 days after surgery
  Blood sample analysis
Change in free fatty acid levels | 24 hours pre-surgery up to 7 days after surgery
  Blood sample analysis
Change in triacylglycerides levels | 24 hours pre-surgery up to 7 days after surgery
  Blood sample analysis
Change in low density lipoprotein levels | 24 hours pre-surgery up to 7 days after surgery
  Blood sample analysis
length of hospital stay | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany